CLINICAL TRIAL: NCT00158795
Title: Assess the Safety & Reactogenicity of GSK Biologicals Hib Vaccine Co-administered With Chinese Local DTPw Vaccine When Compared to Chinese Local DTPw Vaccine Administered Alone, in Healthy Infants at 3,4 & 5 Mths of Age
Brief Title: Assess Safety & Reactogenicity of GSK Biologicals' Hib Vaccine Co-administered With or Without Chinese DTPw Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 104124
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Haemophilus Influenzae Type b Disease
MeSH Terms: interventions — Haemophilus influenza type b polysaccharide vaccine-tetanus toxin conjugate

INTERVENTIONS:
Biological: Haemophilus Influenza type b vaccine

SUMMARY:
To assess safety and reactogenicity of GSK Biologicals' Haemophilus influenza type b vaccine co-administered with or without Chinese DTPw vaccine administered alone in healthy infants (3, 4 and 5 months of age)

DETAILED DESCRIPTION:
All subjects will be randomized into two groups. One group will receive DTPw vaccine co-administered with Hib and another group will receive DTPw vaccine alone. A specific follow-up of solicited local and general symptoms after each vaccination. A specific follow-up of unsolicited symptoms after each vaccination. Recording of serious adverse events reported during the study period.

ELIGIBILITY:
Inclusion Criteria:

* A male or female infant between, and including, 11 and 17 weeks of age at the time of the first vaccination.

Exclusion Criteria:

* Planned administration of a vaccine not foreseen by the study protocol during the period starting 30 days before the administration of the first vaccine dose and ending 30 days after the last dose.
* Chronic administration of immunosuppressants or other immune-modifying drugs from birth until administration of first dose of study vaccine.
* Use of any investigational or non-registered product (drug or vaccine) within 30 days preceding the first dose of study vaccine, or planned use during the study period.

Ages: 3 Months to 4 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 454 (Actual)
Dates: Start 2005-01; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Occurrence of solicited symptoms of grade 3 intensity, during the specific follow-up period after vaccination.

SECONDARY OUTCOMES:
- Occurrence of solicited symptoms during the specific follow up period after vaccination.
- Occurrence of unsolicited symptoms during the specific follow up period after vaccination.
- Occurrence of serious adverse events during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Nanning, Guangxi, China